CLINICAL TRIAL: NCT07079072
Title: The Effects of Acupuncture for Lung Cancer-Related Fatigue, a Clinical Trial
Brief Title: Acupuncture for Lung Cancer-Related Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuanjie Sun, Doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-074-KY-01
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: lung cancer; cancer-related fatigue; acupuncture
MeSH Terms: conditions — Lung Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Device: Acupuncture
- sham acupuncture (Sham Comparator)
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Acupuncture — The main acupoints include Guanyuan (CV4), Zhongwan (CV12), Shangyintang (EX-HN3), bilateral Tianshu (ST25), bilateral Zusanli (ST36), bilateral Hegu (LI4), and bilateral Taichong (LR3). The patient adopts a supine position, and after disinfecting the acupoints, sterile cotton pads are affixed to secure needles.
  In the experimental group, filiform needles measuring Φ0.30×40mm are inserted into the skin to a depth of 0.5-1 cun, achieving "De Qi" sensation. Needles are retained for 30 minutes. At each acupoint (except Shangyintang), manual stimulation including lifting, thrusting, twisting, and plucking is performed once every 10 minutes. The participants received 12 acupuncture sessions over a 4-week period, with three sessions per week scheduled every other day.
  Arms: Acupuncture
Device: Sham Comparator — The acupoints are same with those in the experimental group. The patient adopts a supine position, and after disinfecting the acupoints, sterile cotton pads are affixed to secure needles. The control group use dull needles measuring 0.30 × 25 mm, which are inserted vertically through the fixed pad until reaching the skin surface. The needles are gently lifted, twisted, and rotated slightly three times each, without piercing the skin. The needles are retained for 30 minutes, with no manipulation during this period. The participants received 12 sham acupuncture sessions over a 4-week period, with three sessions per week scheduled every other day.
  Arms: sham acupuncture

SUMMARY:
This study aims to evaluate the efficacy and safety of acupuncture in alleviating cancer-related fatigue (CRF) among lung cancer survivors. It addresses the key issue of limited high-quality evidence for acupuncture's effect on CRF by rigorously comparing real acupuncture against a non-penetrating sham needle control in 120 eligible participants. Patients will be centrally randomized (1:1), blinded, and receive 12-session treatment over 4 weeks. Participants will complete treatment and attend follow-up visits up to week 16, and repeatedly complete fatigue (BFI-C, MFI-20), psychological (PHQ-9, GAD-7, FCRI), functional (CWSAS), and sleep (ISI) assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of lung cancer who have completed initial treatment (including surgery, radiotherapy, and/or chemotherapy) at least 8 weeks prior;
* Aged between 18 and 75 years;
* Meet the diagnostic criteria for cancer-related fatigue;
* Estimated to have a survival period of at least 3 months;
* Patients with moderate to severe cancer-related fatigue (the highest fatigue score in the past 24 hours on the Chinese version of the Brief Fatigue Inventory [BFI-C] ≥ 4 points);
* ECOG Performance Status score ranges from 0 to 2 points
* Voluntarily join this study and sign the informed consent form.

Exclusion Criteria:

* Patients experiencing significant fatigue symptoms before being diagnosed with lung cancer;
* Patients with severe anxiety and depression;
* Patients showing notable cognitive impairment or suicidal tendencies;
* Patients with a history of hypothyroidism or chronic fatigue syndrome;
* Patients suffering from moderate to severe anemia, with hemoglobin levels below 90 g/L;
* Patients experiencing severe pain, with a Numeric Rating Scale (NRS) score of 7 or higher;
* Patients with serious sleep disorders;
* Patients with severe malnutrition;
* Patients with seriously diminished physical function;
* Patients who have undergone acupuncture treatment for cancer-related fatigue within the past month;
* Patients with uncontrolled severe underlying conditions, such as heart failure, myocardial infarction, unstable angina, endocrine disorders, gastrointestinal issues, neurological impairments, severe infections, liver and kidney failure, or chronic obstructive pulmonary disease;
* Patients with poor adherence;
* Patients who are breastfeeding, pregnant, or planning to conceive within the next four months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients whose score of average fatigue over the past 24 hours decreased by at least 2 points on the Brief Fatigue Inventory-Chinese (BFI-C) compared to baseline. | At the 4th week.
  The severity of fatigue is scored on a scale from 0 to 10, higher scores indicating more severe fatigue.

SECONDARY OUTCOMES:
The proportion of patients whose score of average fatigue over the past 24 hours decreased by at least 2 points on the Brief Fatigue Inventory-Chinese (BFI-C) compared to baseline. | At the 8, 12, 16 weeks.
  The severity of fatigue is scored on a scale from 0 to 10, higher scores indicating more severe fatigue.
The change from baseline in the the average fatigue over the past 24 hours on the Brief Fatigue Inventory-Chinese (BFI-C) compared to baseline. | At the 4, 8, 12, and 16 weeks
  The severity of fatigue is scored on a scale from 0 to 10, higher scores indicating more
The proportion of patients whose score on the most severe fatigue over the past 24 hours decreased by 2 points or more on the Brief Fatigue Inventory-Chinese (BFI-C) compared to baseline. | At 4, 8, 12, 16 weeks.
  The total scores for the highest level of fatigue range from 0 to 10 points, higher scores indicating more severe fatigue.
The change from baseline in the the most severe fatigue over the past 24 hours on the Brief Fatigue Inventory-Chinese (BFI-C) compared to baseline. | At the 4, 8, 12, and 16 weeks
  The severity of fatigue is scored on a scale from 0 to 10, higher scores indicating more severe fatigue.
The changes from baseline of Brief Fatigue Inventory-Chinese (BFI-C) scores on quality of life | At 4, 8, 12, 16 weeks.
  The impact of cancer-related fatigue on patients' quality of life is assessed by BFI-C in daily activities, mood, mobility, work, relationships and interests. The score ranges from 0 to 10, with higher score indicating greater impact.
Changes in the scores of the Multidimensional Fatigue Inventory (MFI-20) and the scores of each item compared to the baseline | At 4, 8, 12, 16 weeks.
  Each item scores from 1 to 5 points, the total score ranging from 20 to 100 points, higher scores indicating more severe fatigue.
Changes in the scores of the Fear of Cancer Recurrence Inventory (FCRI ) compared to the baseline | At 4, 8, 12, 16 weeks.
  Each item scores from 0 to 4 points, the total score ranging from 0 to 36 points, higher scores indicating more fear.
Changes in the scores of the Chinese work and social adjustment scale (CWSAS) compared to the baseline | At 4, 8, 12, 16 weeks.
  Each item scores from 0 to 8 points, the total score ranging from 0 to 40 points, higher scores indicating more fear.
Changes in the scores of the Patient Health Questionnaire-9 (PHQ-9) compared to the baseline | At 4, 8, 12, 16 weeks.
  The total score range is 0-27 points, higher scores indicates more severe depression.
Changes in the scores of the Generalized Anxiety Disorder-7 (GAD-7) compared to the baseline | At 4, 8, 12, 16 weeks.
  The total score range is 0-21 points, higher scores indicates more severe anxiety.
Changes in the scores of the Insomnia Severity Index (ISI) compared to the baseline | At 4, 8, 12, 16 weeks.
  The total score range is 0-28 points, higher scores indicates worse results.
The percentage of patients who experienced moderate or significant improvement in fatigue, as evaluated by the Patient Global Impression-Improvement (PGI-I) scale. | At 4, 16 weeks.
  The PGI-I is a patient-reported subjective assessment of their condition, consisting of seven levels: markedly worse, somewhat worse, moderately worse, no change, slightly improved, moderately improved, and markedly improved. The proportion of patients who report moderately improved or markedly improved will be calculated.
Adverse event | From enrollment to the end of follow-up at 16 weeks
  Collect adverse events occurring during treatment and follow-up periods, including acupuncture-related adverse events and other adverse events classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Adherence assessment | From enrollment to the end of follow-up at 16 weeks
  The proportion of subjects who completed 80% or more of acupuncture treatments.
Concomitant medication | From enrollment to the end of follow-up at 16 weeks
  The proportion of patients taking other medications and treatment that could influence fatigue treatment results.

OTHER OUTCOMES:
Assessment of patient's expected benefit from acupuncture treatment | At 0 week.
  Ask the patient, "How do you expect your fatigue to be after four weeks?" Choose from the following options: significantly improved, improved, unsure, unchanged, or worsened.
Assessment of belief in acupuncture | At 0, 4, 16 week.
  Ask the patient, "Do you believe that acupuncture therapy helps in managing your fatigue? " Choose from the following options: ineffective, not very effective, uncertain, somewhat effective, highly effective.
Blinding assessment | Assessment occurs within 5 minutes after the final acupuncture session of any treatment in the last week.
  Ask the patient, "The treatment you received over the past 4 weeks was tradition acupuncture or not?"

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified participant data and data dictionary will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.